CLINICAL TRIAL: NCT04690491
Title: Effect of Menstrual Cyclus Phases of Menstrual Cyclus Phases and Postoperative Pain in Patients With Gynecological Laparoscopy
Brief Title: Mü-opioid Receptor Level and Postoperative Pain in Patients With Gynecological Laparoscopy
Status: Completed | Type: Observational
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Ökkeş Hakan Miniksar, Assistant Professor, Bozok University
Other Study IDs: 189_2019.12.11_07
Record Dates: First submitted 2020-12-22; First posted 2020-12-30 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Gynecological; Surgery (Previous), Affecting Fetus; Postoperative Pain
Keywords: Mu-opioid receptor; Gynecological laparoscopic operation; menstrual cycle
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: follicular cyclus — Days of cyclus 6-12
Other: luteal cyclus — Days of cyclus 20-24

SUMMARY:
The hypothesis that gonadal hormones may affect the perception of pain is an interesting research area.

This prospective observational study will undergo elective laparoscopic gynecological surgery to 18-65 years, is planned to participate in ASA 1-3, 60 volunteer patients.

Patients who have known psychiatric disease and drug-users, an important cardiovascular or central nervous system disease, patients with pain syndromes or routinely using opioid, are non-irregular and predictable cycles of menstrual cycles and very urgent patients will not be included in the study.

In our study, we aimed to determine the relationship between menstrual cyclus phases (follicular and luteal) of menstrual cyclus phases (follicular and luteal) in patients to undergo gynecological laparoscopic operation and the relationship between postoperative pain and opioid analgesic consumption.

DETAILED DESCRIPTION:
This prospective observational study is planned to include 60 volunteer patients aged 18-45, ASA 1-3, undergoing elective laparoscopic gynecological surgery. With the information to be obtained from the patients whose menstrual cycle regularly lasts 21-35 days, the cycle duration will be determined by counting from the first day of the last mens period. Days 6-12 of the cycle will be grouped as follicular (F), and 20-24 as luteal (L). No surgery will be planned during the mens period (1-5 days). Patients will be excluded on days 13-19 of the cycle to better define the two stages.

Remaining 3 ml of blood from routine venous blood samples taken from patients for preoperative evaluation will be stored to investigate μ-Opioid receptor levels. A continuous 10 cm visual analog scale (VAS) will be used to determine the level of postoperative pain.

Researchers who will make postoperative evaluations will be blind to menstrual cycles.

The sensation of pain will be assessed every 10 minutes in the recovery room, intervening with a bolus of 10 mg iv tramadol for a pain score of 3 to 5 and a bolus of 20 mg for a pain score of more than 5. If the VAS does not drop below 3 after two additional tramadol boluses, rescue analgesia will be provided with 2 mg iv morphine.

Patients will be followed in the ward and observations will be made at 6, 12 and 24 hours.

Patients will be asked to evaluate their resting and coughing pains.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer,
* Between the Ages of 18-45,
* Least Primary School Graduate,
* Not Using Drugs That May Affect Cognitive Functions,
* Non-Alcohol Substance Use,
* Patients Without Psychiatric and Neurological Disease.
* Those with regular and predictable menstrual cycles

Exclusion Criteria:

* Those with known psychiatric disease and drugs,
* Those with an important cardiovascular or central nervous system disease,
* Patients with pain syndromes or routinely using opioid,
* Those whose menstrual cycles last less than 21 days and do not have an irregular and predictable menstrual cycle
* Very urgent patients

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Volunteer patients to undergo elective laparoscopic gynecological surgery by the Department of Obstetrics and Gynecology
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-02 (Actual)

PRIMARY OUTCOMES:
Difference between mu opioid receptor levels in menstrual cycle phases | 6 months

SECONDARY OUTCOMES:
Correlation between mu opioid receptor levels and postoperative pain | 6 months
  Correlation between mu opioid receptor levels and postoperative pain

CONTACTS AND LOCATIONS:
Overall Officials: Ökkeş Miniksar, Asist.Prof, Study Chair — YOZGAT BOZOK UNIVERSITY
Locations (1):
- Bozok University Medical Center, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miniksar OH, Onat T, Gocmen AY, Honca M. Serum levels of mu-opioid receptor according to menstrual cycle phases are associated with postoperative pain and opioid consumption in laparoscopic gynecological surgeries: a prospective observational study. Ir J Med Sci. 2023 Aug;192(4):1847-1854. doi: 10.1007/s11845-022-03146-z. Epub 2022 Sep 12. PMID 36094733